CLINICAL TRIAL: NCT06144346
Title: Role of Metastases Directed Radiotherapy in Addition to Standard of Care Systemic Treatment in the Management of Extracranial Oligometastatic Breast Cancer
Brief Title: Metastases Directed Therapy for Oligometastatic Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Rimoun Ramsis Anis Boutrus, Assistant Professor, Radiation Oncology, National Cancer Institute, Egypt
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RO2309-308-080
Record Dates: First submitted 2023-11-04; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Metastatic Cancer; Metastatic Breast Cancer
Keywords: stereotactic radiation; oligometastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Active Comparator): systemic and palliative treatment according to physician discretion
  Interventions: Other: Standard of Care
- Metastases Directed Therapy (Experimental): SABR for all metastatic sites followed by systemic treatment for 6 months
  Interventions: Radiation: Stereotactic Ablative Radiation Therapy
- Locoregional Treatment of the Primary (Experimental): patients who respond to MDT and ST will be randomized to undergo loco-regional treatment or not
  Interventions: Procedure: Locoregional treatment

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiation Therapy — SABR to all metastatic lesions
  Arms: Metastases Directed Therapy
Procedure: Locoregional treatment — mastectomy or BCS for the primary tumor
  Arms: Locoregional Treatment of the Primary
Other: Standard of Care — Systemic treatment and palliative treatment
  Arms: Standard of Care

SUMMARY:
This is a phase III randomized study evaluating the benefit from adding metastases directed therapy and locoregional treatment of the primary in breast cancer patients diagnosed with de novo oligometastatic disease patients will be randomized to receive the standard of care (SOC) treatment vs. systemic treatment + Stereotactic Ablative Radiation Therapy. Responders will be randomized to either undergo loco-regional management of the primary tumor or not

DETAILED DESCRIPTION:
Objectives:

Primary objectives:

• Assessment of the outcome (progression free survival) of patients with extracranial oligometastatic breast cancer receiving standard of care systemic treatment compared to patients receiving ablative radiotherapy in addition to systemic treatment

Secondary objectives:

* Improving quality of life of patients with oligometastatic breast cancer (OMBC)
* Ensuring a safe toxicity profile among the patients receiving SBRT to the metastatic sites in addition to SOC treatment vs patients who receive SOC treatment alone.

Study Methodology:

1. Study Design: Randomized Controlled Trial.
2. Study population & disease Condition: Adult female patients, with pathologically and radiologically proven Oligometastatic breast cancer presenting to National Cancer Institute, Cairo University.
3. Background and Demographic characteristics:

   Adult (>18 years old), Egyptian female patients, who present for treatment in the National Cancer Institute, Cairo University. A detailed informed consent will be signed, proper contraception is a must during systemic and radiotherapy treatment.
4. Inclusion criteria:

i) Female patients aged 18 to 70 years. ii) Pathological evidence of breast cancer, any grade, any T stage. iii) Radiological (at least) evidence of metastatic activity with maximum number of 5 extracranial lesions.

iv) Performance status ≤ 2 v) No pre-existing conditions that may prohibit radiotherapy. e) Exclusion criteria i) Pregnant and lactating women. ii) Prior radiotherapy to affected site(s) in less than a year. iii) Active Connective tissue diseases (e.g Rheumatoid Arthritis). iv) Progression to widespread metastatic disease. v) Cases with brain metastasis

f) Interventions (in details):

Pre-treatment evaluation:

Laboratory studies:

CBC, Liver and Kidney functions and Tumor markers (CA15-3, CEA and CA-125)

Imaging Studies:

Initial Sono-mammography for assessment of local disease (MRI breast to be done whenever indicated, e.g., young patients with dense breast tissue: ACR C&D).

Metastatic workup for establishing oligometastatic status: CT chest, abdomen and pelvis with contrast with Bone scan or PET/CT, more sophisticated imaging techniques to be done in case of failure of modalities to establish the metastatic status (e.g., Dynamic MRI of liver in cases which conventional imaging fails to confirm the nature of a suspected hepatic focal lesion).

Pathological diagnosis: Tru-Cut, core-cut or excisional biopsy from suspicious primary breast mass, also core biopsy from suspected metastatic site whenever indicated.

Treatment plan:

Patients will be randomized into 2 arms: (FIG.A) i) Arm A (interventional) ii) Arm B (control)

* The interventional arm will receive Metastasis Directed Therapy (MDT) using Stereotactic body radiotherapy (SBRT) to oligometastatic lesions initially along with standard of care systemic treatment (SOC) according to discretion of multi-disciplinary team decision.
* The control arm will receive SOC alone.
* Locoregional control to the primary will be done in cases with regressive disease or complete response according to RECIST 1.1 criteria.

The radiation schedule in Arm A will be as follows:

SBRT is recommended to be completed within no more than 3 weeks since the start of the first session. Not all metastases need to receive radiotherapy in the same day, IGRT assisted treatment is a must, PTV expansion will be decided separately for each site treated.

Patients will receive single fraction, 3 fractions or 5 fractions of SBRT according to treated site as follows (Data from NRG BR-002 protocol and ASTRO 2022 conference):

Bone (Peripheral and spine): 18-24Gy/S.S or 30Gy/3fx or 35Gy/5fx Liver: 45-60Gy/3fx or 40-60Gy/5fx Lung: 50-60Gy/3fx (rib tolerance must be met) or 50-60Gy/5fx Others (e.g Adrenals and lymph nodes): according to risk organ tolerances, usually 30Gy/3Fx or 40-60Gy/5fx

Treatment Setup and simulation:

All patients will undergo CT-based treatment planning in with proper immobilization and comfortable setup position. High resolution CT scans should be obtained with uniform slice thickness of ≤ 3mm. When treating multiple metastases such as a lung and extremities, varying the treatment position may be necessary (i.e., simulation with arms up and arms to the side. The use of IV contrast will be required for liver and nodal metastases. For other metastases (central & peripheral lung, cervical/mediastinal, abdominal-pelvic, and spinal/paraspinal), the use of IV contrast is encouraged but will be left to the discretion of the treating physician. As an SBRT protocol, this study requires the use of IGRT, cone-beam CT (CBCT) using a specially mounted kV imaging will be the routine verification method.

Delineation of target volume and organs at risk (OARs):

It will be done using the RTOG contouring guidelines, a maximum intensity projection (MIP) volume will be created in lesion situated in organs with remarkable internal motion (e.g lung lesions), fusion with diagnostic imaging such as PET/CT will be done when delineation of gross lesions is infeasible.

Treatment planning:

General guidelines include the following:

* Multiple coplanar or non-coplanar beam arrangements are acceptable.
* A minimum field dimension of 3 cm should be observed while treating small metastases.
* Doses higher than the prescription isodose (i.e., hotspots) should be manipulated to occur within the target.

Planning SBRT Near Prior Radiotherapy Volumes with toxicity of delivering SBRT to multiple metastases in close proximity to previously irradiated volumes is a bit challenging. A multicenter analysis by German Society of Radiation Oncology (DEGRO) was done in 2021, included patients with primary and secondary pulmonary tumors that has been subject to reirradiation using SBRT to same or near target volumes. It showed feasibility of reirradiation and safe toxicity profile, close adherence to dose constraints made by AAPM TG-101 report will be ensured. Re-irradiated volumes will be delineated with the best possible simulation setup and reproducibility, plans of previous treatment will be fused with overlapping volumes to be minimized as much as possible.

Contouring of Normal Tissue Structures In order to verify each of these limits:

The organs must be contoured such that appropriate volume histograms can be generated.

Dose Tolerance to OARs: will be followed as the SABR consortium guidelines published in 2019.

Data Collection:

Demographic data: Age, family history, comorbidity, grade, stage

Pretreatment Evaluation:

Laboratory, Radiological and pathological data as previously mentioned.

Response Evaluation: by physical examination and standard imaging (CT Chest, abdomen and pelvis with contrast and Bone scan or PET/CT, other specific techniques can be used when indicated), it will follow RECIST 1.1 criteria.

Fig: Consort Diagram showing roadmap of treatment and randomization g) Possible Risk: Acute radiation therapy adverse events will be scored according to the RTOG acute radiation morbidity criteria which is the most commonly used in routine practice.

(Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30; 31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. PMID: 7713792.) Late effects will be reported as per Common Terminology Criteria for Adverse events (CTCAE v5.0) https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm#ctc_50 Adverse events related to SBRT for the treatment of metastases are dependent on the location of the metastases treated, as well as from exposure of surrounding normal tissues. For all treated metastases, fatigue is likely to occur and should be transient, lasting < 8 weeks. Other adverse events are likely to be related to the specific metastatic location receiving SBRT such as esophagitis and pneumonitis during treatment of lung lesions, erythema and alopecia in treatment of bony sites and gastrointestinal upset in volumes related to digestive tract.

Complications of systemic treatment: they shall be discussed in the Multidisciplinary team meeting prior to enrollment in the treatment protocol, patients are also required to be informed about them, the informed consent form for inclusion in this study will have a special section to state the possible side effects of the given systemic treatment as well as radiotherapy.

h) Primary outcome parameters:

* Progression Free Survival (PFS) and Overall Response Rate (ORR) i) Secondary outcome parameters:
* Overall survival (OS)
* Quality of life measurements (QoL) among patients of both arms during the follow up period using Breast Cancer Treatment Outcome Scale (BCTOS) verified questionnaire.
* Occurrence and degrees of treatment related toxicities among patients of both arms during the follow up period.

  j) Sample size: This study aiming to assess progression free survival of patients with extracranial oligometastatic breast cancer receiving either standard of care systemic treatment or ablative radiotherapy in addition to standard of care systemic treatment, with ratio 1:1. Based on previous studies; Glemarec G et al. (2023) & Trovo M et al., (2018), 1 year progression free survival was 93%&75% for systemic treatment alone (group1) and local ablative treatment (group 2) respectively, so we need to study 70 patients per group. This number will be compensated by 5% for suspected losses so the final sample size will be 75 patients per group (total 150 breast cancer patients) to be able to reject the null hypothesis. The Type I error probability associated with test of this null hypothesis is 0.05 & type Ц error was 0.2. Sample size was calculated using Med calc statistical package version (18.2.1) (34, 35).

  k) Statistical analysis: Data management and analysis will be performed using Statistical Package for Social Sciences (SPSS) vs. 28. Numerical data will be summarized using means and standard deviations or medians and ranges, as appropriate. Categorical data will be summarized as numbers and percentages. Numerical data will be explored for normality using Kolmogrov-Smirnov test and Shapiro-Wilk test. Comparisons between two groups for normally distributed numeric variables will be done using the Student's t-test while for non-normally distributed numeric variables, comparisons will be done by Mann-Whitney test. Chi square or Fisher's tests will be used to compare between the groups with respect to categorical data, as appropriate.

Kaplan-meire method will be used to estimate the overall survival and progression free survival. Overall survival will be calculated from date of diagnosis to date of death or last follow up. While progression free survival will be calculated from the date of intiation of treatment to date of progression. Differences between the survival curves will be assessed for statistical significance with the log-rank test. Cox regression analysis will be done to evaluate independent prognostic variables affecting survival time. All tests will be two-sided. P-values < 0.05 will be considered significant.

10-Time plan (when to start/when expected to finish/when to publish) Start from: April 2023 Expected time to finish: March 2025 Expected date for publishing: October 2025 11-Ethical committee approval:

* This study will be started after approval of Institutional Review Board and Ethical Research Committee.
* The study protocol will be presented to the Scientific Ethics Committee of the radiotherapy Department at the National Cancer Institute - Cairo University.
* Patients' data will be presented anonymously with protection of privacy and confidentiality.
* The aim and nature of the study will be explained to each patient before their inclusion in the study. An informed written consent will be obtained from each patient, or a first degree relative before enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 70 years.
* Pathological evidence of breast cancer, any grade, any T stage.
* Radiological (at least) evidence of metastatic activity with maximum number of 5 extracranial lesions.
* Performance status ≤ 2
* No pre-existing conditions that may prohibit radiotherapy.

Exclusion Criteria:

•.Pregnant and lactating women.

* Prior radiotherapy to affected site(s) in less than a year.
* Active Connective tissue diseases (e.g Rheumatoid Arthritis).
* Progression to widespread metastatic disease
* Cases with brain metastasis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological identity
Enrollment: 150 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-08-19 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | from the time of randomization till disease progression or death up-to 120 months
  Time till disease progression
Overall Response rate | assessed using physical exam and PET CT after six months of systemic treatment
  rate of patients responding to therapy

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt